CLINICAL TRIAL: NCT00538577
Title: Outcome and Related Factors of Necrotizing Fasciitis of the Limb
Status: Completed | Type: Observational
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Chacellor of Research, Tehran University of Medical Sciences
Other Study IDs: 86-03-30-6110
Record Dates: First submitted 2007-09-30; First posted 2007-10-02 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Necrotizing Fasciitis
Keywords: Necrotizing fasciitis
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Soft tissue necrotizing fasciitis of limbs are lethal infections and associated with high morbidity and mortality rates. The purpose of this study is to determine the clinical manifestations and factors affected the treatment outcome to predict the prognosis and make timely decision for appropriate management and prevent limb loss.

DETAILED DESCRIPTION:
Patients that are admitted to hospital with the diagnosis of necrotizing fasciitis of a limb will be entered to this study. A questionnaire will be completed for each patient included demographic data, admission and diagnosis date, treatment onset, medical history for diabetes mellitus, HIV infection, use of immunosuppressor drugs, peripheral vascular disease, cancer, renal disease, intravenous drug abuse, and disease outcome that can be recovery, amputation or death.

ELIGIBILITY:
Inclusion Criteria:

* Necrotizing fasciitis of the limb

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Patients with diagnosis of necrotiying faciitis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Espandar, MD, Principal Investigator — Imam Khomeini Hospital- Tehran University of Medical Sciences
Locations (1):
- Operative Theater of Orthopedic Surgery Department- Imam Khomeini Hospital, Tehran, Tehran Province, Iran